CLINICAL TRIAL: NCT01988948
Title: Impact de la Vaccination Sur la Distribution Des génotypes de Papillomavirus (HPV) et Suivi de la Dynamique Intra-individuelle de l'Infection et Des Co-infections Dans Une Population d'étudiantes âgées de 18 à 20 Ans
Brief Title: Dynamics of Human PApilloma Virus Interactions; Internet-based Students HeAlth Research Enterprise
Acronym: DyPAVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Versailles Saint-Quentin-en-Yvelines University (Other); centre national de référence pour les Papillomavirus Humains (Unknown); German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-42; 2012-A00814-39 (Other: ID-RCB)
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Infection by Human Papilloma Virus
Keywords: Human papilloma virus; Young women; I-Share

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- student cohort (Other): Various biological sampling
  * blood sampling,
  * oral, vulvar, vaginal and anal sampling for women,
  * oral and genital sampling for men
  Interventions: Other: Various biological sampling

INTERVENTIONS:
Other: Various biological sampling

SUMMARY:
Human papillomavirus (HPV) infection is the most common sexually transmitted infection. The high risk oncogenic types, HPV-16 and -18 are responsible for 70% of cervical cancers. The introduction of vaccination against two major oncogenic genotypes of HPV raises questions about genotype replacement because of the existence of other oncogenic types not targeted by the vaccine. A better understanding of natural history of HPV infection and interaction (competition, synergy) between genotypes are required in order to anticipate this phenomenon.

The aims of this study are to characterize HPV infection in young female students and to follow up HPV infection and co-infection dynamics with different genotypes, taking into account both vaccination status and immunity to HPV 16 and 18. The study also focuses on the determination of factors influencing the development of persistent cervical HPV infections.

The DyPAVIR-ISHARE study is based on the participation of 5000 young female students, from 18 to 20 years-old, all registered at the Universities of Bordeaux or Versailles Saint-Quentin (UVSQ). The 3-years follow-up includes completion of a self-administrated questionnaire regarding sexual behaviour, socio-demographic characteristics, access to health-care services and, for a sub-group of 1000 students, the taking of genital and oral self-taken samples for the detection and genotyping of HPV (every 3 months). Previously, a pilot phase study (2 visits in 3 months of interval) is set up on 50 young female students from UVSQ in order to test feasibility.

This study will provide data to gain insight into the possibility of type replacement. Moreover, this study would provide an overview of HPV vaccine coverage and effectiveness HPV incidence and factors associated with HPV infection and co-infection ; Partners recruitment would allow us to follow HPV transmission dynamics among couples, and in particular, HPV exposure in young adult women. The HPV research won't be limited to virus detection in samples but will indicate the presence or absence of HPV infection.

Finally, additional genetic studies could be conducted in order to study genetic susceptibility to HPV infection, to chronic HPV infection and to co-infection.

This research project is part of the i-Share program funded by the "Investissement d'Avenir" cohort call.

ELIGIBILITY:
Women

Inclusion Criteria:

* voluntary student consulting the health service of university
* age 18-20 y.o.
* informed consent signed
* affiliated to national health insurance

Exclusion Criteria:

* pregnancy
* end of the pregnancy within the last 3 months
* Student participating in another clinical trial

Men

Inclusion Criteria:

* being the sexual partner of a woman included in this study
* at least 18 y.o
* informed consent signed
* affiliated to national health insurance

Exclusion Criteria:

none

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of HPV detection at inclusion (all HPV genotypes) | 2 years

SECONDARY OUTCOMES:
Incidence of oncogenic HPV genotypes, co-infection with different HPV genotypes | 5 years

OTHER OUTCOMES:
Factors associated with HPV infection and co-infection | 5 years
HPV clearance (all genotypes and genotype-specific HPV) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Didier Guillemot, Pr, MD, Study Director — Unité Pharmacoépidémiologie et maladies infectieuses (PhEMI), Institut Pasteur / Université Versailles Saint-Quentin-en-Yvelines / INSERM; Elisabeth Delarocque-Astagneau, MD, Study Director — Unité Pharmacoépidémiologie et maladies infectieuses (PhEMI), Institut Pasteur / UVSQ / Inserm; Emmanuelle Mathiot-Vicaigne, MD, Principal Investigator — Versailles Saint-Quentin-en-Yvelines University
Locations (1):
- Service Universitaire de Médecine Préventive et de Promotion de la Santé (SUMPPS), Versailles, France

IPD SHARING:
Plan to Share IPD: Undecided